CLINICAL TRIAL: NCT01095900
Title: Comparison of Botulinum Toxin and Sphincterotomy in the Treatment of Chronic Anal Fissure
Status: Completed | Type: Observational
Sponsor: Theodor Bilharz Research Institute (Other)
Other Study IDs: TheodorBRI
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Pain
Keywords: Pain after treatment; healing of fissure after treatment; continence scores after treatment
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- LIS group)
  Interventions: Procedure: conservative lateral internal sphincterotomy
- BT group
  Interventions: Procedure: Intra-sphincteric Botulinum-toxin injection

INTERVENTIONS:
Procedure: conservative lateral internal sphincterotomy
  Groups: LIS group)
Procedure: Intra-sphincteric Botulinum-toxin injection
  Groups: BT group

SUMMARY:
Intra-sphincteric injection of botulinum toxin seems to be a reliable option causing temporary alleviation of sphincter spasm and allowing the fissure to heal. study is to compare the outcome of surgical sphincterotomy and botulinum toxin injection treatments in patients with uncomplicated chronic anal fissure.

DETAILED DESCRIPTION:
consecutive patients with uncomplicated chronic anal fissure who had failed conservative treatment were randomized to receive either intra-sphincteric injection of botulinum toxin (BT) or lateral internal sphincterotomy (LIS). Postoperative pain relief, healing of fissure, continence scores and fissure relapse during 18 weeks of follow up was the outcomes assessed.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of chronic anal fissure was based on evidence of circumscribed ulcer at anal canal with indurations at the edges and exposure of the horizontal fibers of the internal anal sphincter at its floor.

Exclusion Criteria:

* Anal fissure that had been operated on before, complicated fissure with cicatricial deformation, large sentinel pile, associated hemorrhoids, suspected inflammatory bowel disease, or malignancy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This trial included consecutive adult patients presenting with symptomatic chronic anal fissure in which conservative treatment had failed.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain relief, healing of fissure, continence scores | 18 weeks

SECONDARY OUTCOMES:
fissure relapse | 18 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery-Theodore Bilharz Research Institute ,, Cairo, Egypt